CLINICAL TRIAL: NCT05978687
Title: The Use of Lidocaine Ophtesic Gel Versus Subconjunctival Xylocaine Injection in Pterygium Excision
Brief Title: The Use of Lidocaine Gel Versus Subconjunctival Xylocaine Injection in Pterygium Excision
Acronym: LIDPTER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Karolien Termote, MD FEBOpht, Ophthalmologist, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23149_Pterygium
Record Dates: First submitted 2023-07-03; First posted 2023-08-07 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Pterygium
Keywords: Lidocaine gel; Pterygium; Dryness; Irritation
MeSH Terms: conditions — Pterygium | interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical lidocaine gel (Experimental): All patients will receive topical 2% lidocaine gel (Ophtesic lidocaine gel) prior to surgery
  Interventions: Drug: OPHTESIC LIDOCAINE HYDROCHLORIDE 20MG/G
- Subconjunctival xylocaine injection (Active Comparator): All patients will receive a subconjunctival injection with xylocaine 2% hydrochloride solution with 0.125 epinephrine will be injected with a 27-gauge needle
  Interventions: Drug: Xylocaine with Epinephrine

INTERVENTIONS:
Drug: OPHTESIC LIDOCAINE HYDROCHLORIDE 20MG/G — In group A, all patients will receive topical 2% lidocaine gel (ophtesic lidocaine hydrochloride 20 mg/G) prior to surgery.
  Operative technique A traction suture is applied at the superior limbus (Vicryl 6.0) with a Kocher. The head of the pterygium is separated from its body with scissors. Afterwards it is removed by blunt dissection. The subconjunctival tissue under the body of the lesion is removed. The conjunctival graft is separated from the Tenon's capsule for harvest by ballooning with SBSS in group A and by injection with 0.5 mL of 2% xylocaine in group B. The autograft is excised from the superior temporal side. Hereafter, the graft is secured to the recipient bed with sutures. The traction suture is removed. All operations are executed by the same surgeon.
  Other Names: Lidocain gel
  Arms: Topical lidocaine gel
Drug: Xylocaine with Epinephrine — In group B, all patients will receive a subconjunctival injection with xylocaine 2% hydrochloride solution with 0.125 epinephrine will be injected with a 27-gauge needle. When asked for, patients will receive additional topical 1% lidocaine eye drops.
  Operative technique A traction suture is applied at the superior limbus (Vicryl 6.0) with a Kocher. The head of the pterygium is separated from its body with scissors. Afterwards it is removed by blunt dissection. The subconjunctival tissue under the body of the lesion is removed. The conjunctival graft is separated from the Tenon's capsule for harvest by ballooning with SBSS in group A and by injection with 0.5 mL of 2% xylocaine in group B. The autograft is excised from the superior temporal side. Hereafter, the graft is secured to the recipient bed with sutures. The traction suture is removed. All operations are executed by the same surgeon.
  Other Names: Subconjucntival injection with xylocain injection
  Arms: Subconjunctival xylocaine injection

SUMMARY:
In pterygium excision procedures, the subconjunctival injection of xylocain is regarded as an uncomfortable and painful step in the procedure. While already being studied in other ophthalmic procedures such as glaucoma surgery (7), application of topical lidocaine gel is likely to minimize pain. The gel has a longer surface contact time due to its consistency, providing not only a longer anesthetic effect, but protecting the corneal surface against desiccation, when compared to eye drops.

The investigators hypothesize that Ophtesic 2% lidocaine gel is as effective as an anesthetic in pterygium excision as subconjunctival injection, while providing more comfort during surgery and less corneal dryness afterwards.

Our goal is to compare both the anesthetic and corneal surface effect of topical 2% lidocaine gel to subconjunctival injection of xylocaine 2% solution with 0.125 epinephrine in pterygium surgery:

* Compare the patients pain during and after surgery
* Compare corneal dryness after surgery.
* Evaluate possible secondary events

DETAILED DESCRIPTION:
Pterygia are known as fibrovascular degenerations in the outer layer of the eye. Usually, they cross the limbus onto the cornea. they develop over time and can cause symptoms such as redness, itching, irritation and decreased vision. In severe cases, pterygia can provoke binocular diplopia due to contraction of the Tenon's capsule. Risk factors are age, UV exposure and male gender.

Rezvan F. et al conducted a meta-analysis to study the prevalance of pterygia in the world. Their prevalence is estimated at 12% in the worldwide population, being higher in subtropical regions. They occur slightly more in men, 13% versus 12%, when compared to women. The highest prevalence is seen in patients over 80 years old (up to 19.5%).

The exact mechanism of pathogenesis is not clear. A pterygium consists of degenerated collagen tissue. Several previous studies have already proven the role of anti-apoptotic proteins such as p53, a tumor suppressor protein. Its expression is elevated when compared to normal conjunctival tissue. UV exposure is the most important risk factor. This theory is supported by histopathologic actinic changes, similar to actinic keratosis, seen in pterygia.

First line treatment for pterygia are conservative measures, like lubricants and sunglasses to protect against additional harmful UV radiation. Yet, these measures are only symptomatic and will not eliminate the cause. Surgery is regarded as an ideal solution in patients who would like a definitive improvement of esthetic and visual problems. Several surgery techniques are already known, but the most common is closure of the excised pterygium with a conjunctival auto graft. In this technique, conjunctiva from the superotemporal limbal part of the patient's eye is used to cover the excised pterygium area. A systematic review compared the risk of recurrence of this technique to the use of an amniotic membrane and concluded that the risk of recurrence was 46% percent less in the first group.

These days, subconjunctival injection of xylocaine 2% solution with 0.125 epinephrine is the most used anesthesia technique. The anesthesia is infero- or superotemporal administered 5-8mm from the limbus. While giving excellent anesthetic result, the pain and anxiety caused by this injection implied the need for new techniques. In chalazion and cataract surgery, lidocaine gel is already confirmed to have a sufficient anesthetic effect on patients while the amount of pain and anxiety during administration was decreased. In pterygium surgery, both and proves that pain was less during both anesthesia administration and post-operatively. Now that Ophtesic lidocaine gel is also on-label for pterygium excision, in many centers the gel is used as standard of care.

With Oksuz et al. (3) already having investigated the efficacy of lidocaine gel in pterygium surgery, there might be more advantages yet to be investigated. For example, the lidocaine gel has the advantage of having a viscous consistency. This allows the gel to protect the eye from desiccating during surgery. Our primary goal in this study is to compare the ef-fect on dryness and irritation in patients after pterygium surgery with both methods of an-aesthesia by using the OSDI score questionnaire and the Oxford Dry Scale. In addition to equal anaesthetic effect, this could push the standard of care in favour of the lidocaine gel.

In pterygium excision procedures, the subconjunctival injection of xylocaine is regarded as an uncomfortable and painful step in the procedure. Already proved to be equal, the gel has a longer surface contact time due to its consistency, providing not only a longer anesthetic effect, but protecting the corneal surface against desiccation, when compared to eye drops. Nowadays, it is already considered as the standard of care.

The investigators hypothesize that Ophtesic 2% lidocaine gel is as effective as an anesthetic in pterygium excision as subconjunctival injection, while providing more comfort during surgery and less corneal dryness afterwards.

Our goal is to compare both the anesthetic and corneal surface effect of topical 2% lidocaine gel to subconjunctival injection of xylocaine 2% solution with 0.125 epinephrine in pterygium surgery:

* Compare the patients pain during and after surgery
* Compare corneal dryness after surgery.
* Evaluate possible secondary events (e.g. enophtalmitis or non-adherence of the graft)

Procedure Anesthesia In group A, all patients will receive topical Povidone- Iodine and 2% lidocaine gel prior to surgery. In group B, all patients will receive Povidone- Iodine and a subconjunctival injection with xylocaine 2% hydrochloride solution with 0.125 epinephrine will be injected with a 27-gauge needle. When asked for, patients will receive additional topical 1% lidocaine eye drops.

Operative technique A traction suture is applied at the superior limbus (Vicryl 6.0) with a Kocher. The head of the pterygium is separated from its body with scissors. Afterwards it is removed by blunt dissection. The subconjunctival tissue under the body of the lesion is removed. The conjunctival graft is separated from the Tenon's capsule for harvest by ballooning with SBSS in group A and by injection with 0.5 mL of 2% xylocaine in group B. The autograft is excised from the superior temporal side. Hereafter, the graft is secured to the recipient bed with sutures. The traction suture is removed. All operations are executed by the same surgeon.

Following outcomes will be assessed:

• Pain The investigators will monitor pain assessment with the Visual Analogue Pain Scale. Patients will be asked to give a score from 0 (no pain at all) to 10 (worst pain imaginable). The assessment is done intra- and post- operatively by a nurse of the department. During both assessments, the surgeon will leave the operating room.

Pain will be monitored at following moments:

* Initial administration of anesthesia
* At incision
* Within 5 minutes after surgery
* Day one post-operative consult

  * Dryness The dryness is assessed in two manners. The Oxford Dry Eye Scale (11) (Figure two) will be handled as an objective tool to grade dryness. The Ocular Surface Disease Index OSDI (12) (Figure three, four and five) is a subjective manner of assessing dryness. The questionnaire will be available in English, Dutch and French.

At following moments the dryness will be monitored:

* Day one post-operative consult
* Day 8 post-operative consult

Exclusion criteria:

* History of auto-immune diseases such as Sjögren, Lupus, Graves, Graft-versus-host disease, rheumatoid arthritis.
* History of deafness, anxiety disorders, communicative barrier, impossibility to comprehend the Visual Analogue Pain Scale or the OSDI questionnaire.
* Patient who already had pterygium excision

ELIGIBILITY:
Inclusion Criteria:

* Indication of pterygium excision

Exclusion Criteria:

* No history of auto-immune diseases such as Sjögren, Lupus, Graves, Graft-versus-host disease, rheumatoid artritis
* No history of deafness, anxiety disorders, communicative barrier, impossibility to comprehend the Visual Analogue Pain Scale or the OSDI questionnaire.
* Patient who already had pterygium excision

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in OSDI score POD8 | Post-op day 8
  The Ocular Surface Disease Index OSDI (12) is a subjective manner of assessing dryness. The questionnaire will be available in English, Dutch and French. Our primary outcome is the difference in OSDI score between both groups after 8 days.

SECONDARY OUTCOMES:
Secondary events | Post-op day 8
  Number of secondary events in absolute numbers (non-adherence of graft, endophtalmitis, ...)
Change of OSDI score | Post-op day 1 to 8
  The Ocular Surface Disease Index OSDI (12) is a subjective manner of assessing dryness. The questionnaire will be available in English, Dutch and French. A secondary outcome is the mean difference of the OSDI score between both groups.
Pain via Visual Analogue Pain Scale at administration of anesthesia | Per-operative at administration of anesthesia
  We will monitor pain assessment with the Visual Analogue Pain Scale. Patients will be asked to give a score from 0 (no pain at all) to 10 (worst pain imaginable).
Pain via Visual Analogue Pain Scale at incision | Per-operative at incision
  We will monitor pain assessment with the Visual Analogue Pain Scale. Patients will be asked to give a score from 0 (no pain at all) to 10 (worst pain imaginable).
Pain via Visual Analogue Pain Scale < 5 minutes after the operation | <5 minutes after operation
  We will monitor pain assessment with the Visual Analogue Pain Scale. Patients will be asked to give a score from 0 (no pain at all) to 10 (worst pain imaginable).
Pain via Visual Analogue Pain Scale 1 day after the operation | Post-op day 1
  We will monitor pain assessment with the Visual Analogue Pain Scale. Patients will be asked to give a score from 0 (no pain at all) to 10 (worst pain imaginable).
Pain via Visual Analogue Pain Scale 8 days after the operation | Post-op day 8
  We will monitor pain assessment with the Visual Analogue Pain Scale. Patients will be asked to give a score from 0 (no pain at all) to 10 (worst pain imaginable).
Change in pain via Visual Analogue Pain Scale | pre-operative, post-op day 1 and day 8
  We will monitor pain assessment with the Visual Analogue Pain Scale. Patients will be asked to give a score from 0 (no pain at all) to 10 (worst pain imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Karolien Termote, Master, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- UZ Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oksuz H, Tamer C. Efficacy of lidocaine 2% gel in pterygium surgery. Acta Ophthalmol Scand. 2005 Apr;83(2):206-9. doi: 10.1111/j.1600-0420.2005.00404.x. PMID 15799734